CLINICAL TRIAL: NCT00391755
Title: A Double-Blind Placebo-Controlled Trial of Rozerem in Migraine Headaches
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit necessary number of patients.
Sponsor: Charlottesville Neuroscience (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Patricia Shipley, MD, Principal Investigator, Charlottesville Neuroscience
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-013R
Record Dates: First submitted 2006-10-22; First posted 2006-10-24 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Migraine Headache
Keywords: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): ramelteon 8 mg po qhs with sleep and migraine journal
  Interventions: Drug: ramelteon
- 2 (Placebo Comparator): Placebo po qhs with sleep and migraine journal
  Interventions: Drug: ramelteon

INTERVENTIONS:
Drug: ramelteon — 1. ramelteon 8mg po qhs with sleep and headache diary
  2. placebo 1 po qhs with sleep and headache diary
  Other Names: Rozerem

SUMMARY:
To study the effect of Rozerem, a high affinity MT1 and MT2, low affinity 5-HT2B receptor agonist used for insomnia, as a migraine prophylactic agent.

DETAILED DESCRIPTION:
In a recent, large study of migraineurs, over half reported difficulties with sleep initiation or maintenance. Those who had shorter average sleep times reported more severe headaches. Poor sleep has been associated with increased frequency and severity of migraines. The improvement of migraine frequency with improved sleep hygiene has been documented.

PET imaging has shown increased regional cerebral blood flow to neural structures involved in the sleep wake cycle during migraine headaches. Polysomnography has shown specific headache types to occur in specific sleep stages.

Melatonin has been effective primarily in headache due to delayed sleep phase syndrome. Recent studies support the efficacy of melatonin in treating migraine. The purpose of this study is to examine the efficacy of Rozerem as a prophylactic migraine medication. If effective, the benefits of the drug as a prophylactic agent for migraine include the tolerability of the drug and the possible secondary benefit of improvement in sleep.

Hypothesis: Rozerem will decrease migraine frequency due to the improvement in sleep and possibly due to the shared neurophysiology of sleep and migraine affected by melatonin.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* 3-8 Migraine headaches/month
* Able to understand and comply with the study

Exclusion Criteria:

* Currently on migraine prophylaxis
* Currently on sleep medication > 4days/month
* Currently on Fluvoxamine
* Untreated psychiatric or sleep disorders
* MRI abnormalities other than those attributable to migraine headaches
* Abnormalities on neurological exam other than known neurological disorders unassociated with migraine or sleep
* Known disorders of prolactin
* Bipolar disorder
* Hepatic disease
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Statistically significant reduction in migraine headaches in the Rozerem treated group. | 4 months

SECONDARY OUTCOMES:
Improvement in sleep satisfaction in the Rozerem treated group. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Shipley, MD, Principal Investigator — Charlottesville Neuroscience
Locations (1):
- Patricia Shipley, MD, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Sahota PK, Dexter JD. Sleep and headache syndromes: a clinical review. Headache. 1990 Jan;30(2):80-4. doi: 10.1111/j.1526-4610.1990.hed3002080.x. PMID 2406223
- [Background] Kelman L, Rains JC. Headache and sleep: examination of sleep patterns and complaints in a large clinical sample of migraineurs. Headache. 2005 Jul-Aug;45(7):904-10. doi: 10.1111/j.1526-4610.2005.05159.x. PMID 15985108
- [Background] Boardman HF, Thomas E, Millson DS, Croft PR. Psychological, sleep, lifestyle, and comorbid associations with headache. Headache. 2005 Jun;45(6):657-69. doi: 10.1111/j.1526-4610.2005.05133.x. PMID 15953298
- [Background] Bruni O, Galli F, Guidetti V. Sleep hygiene and migraine in children and adolescents. Cephalalgia. 1999 Dec;19 Suppl 25:57-9. doi: 10.1177/0333102499019s2516. PMID 10668125
- [Background] Bahra A, Matharu MS, Buchel C, Frackowiak RS, Goadsby PJ. Brainstem activation specific to migraine headache. Lancet. 2001 Mar 31;357(9261):1016-7. doi: 10.1016/s0140-6736(00)04250-1. PMID 11293599
- [Background] Peres MF. Melatonin, the pineal gland and their implications for headache disorders. Cephalalgia. 2005 Jun;25(6):403-11. doi: 10.1111/j.1468-2982.2005.00889.x. PMID 15910564
- [Background] Peres MF, Zukerman E, da Cunha Tanuri F, Moreira FR, Cipolla-Neto J. Melatonin, 3 mg, is effective for migraine prevention. Neurology. 2004 Aug 24;63(4):757. doi: 10.1212/01.wnl.0000134653.35587.24. No abstract available. PMID 15326268